CLINICAL TRIAL: NCT02774109
Title: The Effects of Fish Oil on Patients With Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FishOilonCNLBP201604
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; fish oil; omega 3
MeSH Terms: conditions — Low Back Pain | interventions — Fish Oils; Fatty Acids, Omega-3; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group will take fish oil (five 1000mg fish oil soft capsules per day, each capsule containing 350mg EPA and 250mg DHA) and receive physical modality treatment (hotpacking 15min and transcutaneous electrical nerve stimulation (TENS) 15min, three times a week) for 8 weeks
  Interventions: Dietary Supplement: Fish oil; Procedure: Hotpacking; Procedure: Transcutaneous electrical nerve stimulation (TENS)
- Control group (Placebo Comparator): Participants in the control group will take placebo (five 1000mg sunflower oil soft capsules per day) and receive physical modality treatment (hotpacking 15min and transcutaneous electrical nerve stimulation (TENS) 15min, three times a week) for 8 weeks
  Interventions: Dietary Supplement: Placebo; Procedure: Hotpacking; Procedure: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Dietary Supplement: Fish oil — Five 1000mg fish oil soft capsules per day (each capsule containing 350mg EPA and 250mg DHA) for 8 weeks
  Other Names: omega 3 polyunsaturated fatty acid
  Arms: Experimental group
Dietary Supplement: Placebo — Five 1000mg sunflower oil soft capsules per day for 8 weeks
  Arms: Control group
Procedure: Hotpacking — Hotpacking 15min on low back, three times a week for 8 weeks
Procedure: Transcutaneous electrical nerve stimulation (TENS) — Transcutaneous electrical nerve stimulation (TENS) 15min on low back, three times a week for 8 weeks

SUMMARY:
Objectives:

To investigate the efficacy of omega-3 polyunsaturated fatty acids (PUFA) on patients with chronic nonspecific low back pain (NLBP).

Methods and Materials:

Twenty-nine patients with chronic NLBP were randomly divided into experimental and control groups. For 8 weeks, participants in the experimental group received omega-3 PUFA at 3000 mg/day plus physical therapy, while those in the control group received placebo plus physical therapy. The visual analog pain scale, pressure algometer, Biering-Sorenson test, Roland-Morris Low Back Pain and Disability Questionnaire (RMQ), and occupational burnout inventory (OBI) were used in assessments at baseline (T0) and after 4 (T1) and 8 weeks (T2). Serum erythrocyte sedimentation rate (ESR) and hypersensitive C-reactive protein (hs-CRP) were checked at baseline and T2.

DETAILED DESCRIPTION:
Low back pain is a common symptom in modern society. However, nearly 85% of those who seek medical care for low back pain have no specific history and no specific finding in image study, and therefore do not receive a specific diagnosis. This type of low back pain is termed "nonspecific low back pain." Fish oil contains omega-3 polyunsaturated fatty acid, including eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). EPA and DHA can reduce the synthesis of prostaglandin E2. They are also the precursors of the E-resolvin and D-resolvin that suppress inflammatory cytokine production and act to resolve inflammation. Several previous studies showed that fish oil has the effect of anti-inflammation and pain reduction without side effect that affecting stomach and renal function. Therefore, fish oil is considered a new type of NSAID, and many studies are investigating its effect of anti-inflammation and pain reduction on different diseases. The purpose of this study is to investigate the effects of fish oil on patients with chronic nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 20-50
* Low back pain duration over 3 months and pain intensity over 40mm when assessed with 100mm VAS

Exclusion Criteria:

* History of major trauma or surgery at back
* Obvious spinal pathology on plain film (e.g. scoliosis, spondylosis, spondylolisthesis)
* Not suitable for taking fish oil or receiving physical modality treatment
* Having other inflammatory disease (e.g. rheumatic arthritis, endometriosis, ankylosing spondylitis, infection)
* Pregnancy
* Regularly taking fish oil or fatty fish more than 2 times per week
* Having coagulopathy or currently taking anti-coagulation agent
* Receiving oral or topical NSAID in the past one week
* Taking oral corticosteroid in the past 6 weeks
* Receiving local injection of corticosteroid or prolotherapy in the past 3 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
100mm Visual Analogue Scale (VAS) | Week 8 (T2)
  Assess low back pain intensity (current, least and worst in the past one week)

SECONDARY OUTCOMES:
Pressure pain threshold | Baseline (T0), Week 4 (T1), Week 8 (T2)
  Assess pressure pain threshold with pressure algometer at quadratus lumborum and sacroiliac joint
Roland Morris Low Back Pain and Disability Questionnaire (RMQ) | Baseline (T0), Week 4 (T1), Week 8 (T2)
  Assess the impact of low back pain on daily life with Taiwan version of Roland Morris Low Back Pain and Disability Questionnaire
Biering-Sorenson test | Baseline (T0), Week 4 (T1), Week 8 (T2)
  Assess back extensor endurance
Occupational burnout inventory | Baseline (T0), Week 4 (T1), Week 8 (T2)
  Assess objective occupational burnout feeling
100mm Visual Analogue Scale (VAS) | Baseline (T0), Week 4 (T1)
  Assess low back pain intensity (current, least and worst in the past one week)
Blood test: ESR | Baseline (T0) and Week 8 (T2)
  Draw 10ml blood for checking the level of ESR
Blood test: hs-CRP | Baseline (T0) and Week 8 (T2)
  Draw 10ml blood for checking the level of hs-CRP

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hsun Yang, MD, Principal Investigator — Kaohsiung Chang Cung Memorial Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No